CLINICAL TRIAL: NCT03102788
Title: Task Shifting in the Care for Patients With Hand Osteoarthritis: May the First Consultation in Specialist Health Care be Performed by an Occupational Therapy Specialist?
Brief Title: Task Shifting in the Care for Patients With Hand Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Resource Center for Rehabilitation in Rheumatology (Other)
Collaborators: Diakonhjemmet Hospital (Other); Martina Hansen Hospital (Unknown)
Responsible Party: Principal Investigator, Ingvild Kjeken, Professor, National Resource Center for Rehabilitation in Rheumatology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Project nr 97001
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis Both Hands

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial, participants will be allocated to receive their first consultation in specialist health care by either an occupational therapy specialist or a rheumatologist. The occupational therapist may thereafter refer the patient to a consultation with a rheumatologist if necessary, and vice versa.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research assistant who will examine the participants at baseline and follow-ups and the statistician who perform the main effect analysis will be blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients in the control group will receive their first consultation in specialist health care by a rheumatologist. Rheumatologist-led care comprises confirmation of diagnosis, information about hand osteoarthritis and symptom modifying medication, and, for some patients, Intra-articular injection of long-acting Corticosteroid. The rheumatologist may also refer participants to occupational therapy if needed.
  Interventions: Behavioral: Rheumatologist-led care.
- Intervention (Experimental): Patients in the intervention group will receive their first consultation in specialist health care by an occupational therapy specialist. Occupational therapist-led care comprises confirmation of diagnosis, information about hand osteoarthritis and symptom modifying medication, teaching of hand exercises and ergonomic working methods, and, for some patients, provision assistive devices and orthoses/splints. The occupational therapist will refer patients to a short rheumatologist consultation if confirmation of diagnosis or intra-articular injections of long-acting Corticosteroid are needed.
  Interventions: Behavioral: Occupational therapist-led care.

INTERVENTIONS:
Behavioral: Rheumatologist-led care. — Rheumatologist-led care comprises confirmation of diagnosis, information about hand osteoarthritis and symptom modifying medication, and, for some patients, Intra-articular injection of long-acting Corticosteroid.
  The rheumatologist may also refer participants to occupational therapy if needed.
  Arms: Control
Behavioral: Occupational therapist-led care. — Occupational therapist-led care comprises confirmation of diagnosis, information about hand osteoarthritis and symptom modifying medication, teaching of hand exercises and ergonomic working methods, and, for some patients, provision assistive devices and orthoses/splints. The occupational therapist will refer patients to a short rheumatologist consultation if confirmation of diagnosis or intra-articular injections of long-acting Corticosteroid are needed.
  Arms: Intervention

SUMMARY:
The main aim in this randomized controlled trial is to improve access to safe and effective care, professional practice and cost-effective utilisation of health care resources by testing if occupational therapist-led care is as effective and safe as rheumatologist-led care for people with hand osteoarthritis.

DETAILED DESCRIPTION:
Hand osteoarthritis is one of the most prevalent musculoskeletal conditions in an adult population, and may have large influences on an individual's function, health related quality of life, and participation in the society. In the absence of disease-modifying interventions, occupational therapy, comprising information, hand exercises, assistive devices and orthoses/splints, is considered as core treatment. In Norway, people with hand osteoarthritis are increasingly referred to consultation by a rheumatologist in specialist health care. At the same time a shortage of rheumatologists nationwide is stressing the healthcare system's capacity, and rheumatologists time should therefore primarily be allocated to patients in which early diagnosis and medical treatment are essential.

The World Health Organization recommend task-shifting as one method of strengthening and expanding the health workforce. Such models rely on other healthcare providers in expanded clinical roles, where physiotherapists, nurses or occupational therapists working in collaboration with physicians and other team members have their own patients for whom they provide health care services.

In this randomized controlled trial, we will test if a new model, where patients referred to consultation in specialist health care receive their first consultation by an occupational therapy specialist, is as safe and effective as the traditional model, where they receive their first consultation by a rheumatologist.

ELIGIBILITY:
Inclusion Criteria:

* Hand osteoarthritis diagnosed by physician in primary care, referred for consultation in specialist health care, and ability to communicate in Norwegian.

Exclusion Criteria:

* Exclusion criteria were cognitive or mental impairment, possible inflammatory rheumatic disease (SR>40 or CRP>20, or patient confirming having psoriasis during telephone screening).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Number of treatment responders | One year
  Number of treatment responders will be calculated as number of OMERACT/OARSI-responders. This is a composite index that presents the results of changes after treatment in the three domains of pain, function and patient's global assessment as a single variable (responder yes/no).

SECONDARY OUTCOMES:
Number of painful finger joints | One year
  Joint count of number of painful finger joints at each hand
Hand pain measured on a numeric rating scale | One year
  Hand pain will be measured on a numeric rating scale
Hand stiffness measured on a numeric rating scale | One year
  Hand stiffness will be measured on a numeric rating scale
Disease activity measured on a numeric rating scale | One year
  Disease activity will be measured on a numeric rating scale
Physical function measured by the Functional Index for Hand OsteoArthritis | One year
  Physical function will be measured by the Functional Index for Hand OsteoArthritis
Activity performance measured by the Measure of Activity Performance of the Hand | One year
  Activity performance will be measured by the Measure of Activity Performance of the Hand
Grip strength measured by JAMAR dynamometer | One year
  Grip strength will be measured by JAMAR dynamometer
Health related quality of life measured by EQ5D | One year
  Health related quality of life will be measured by EQ5D
Satisfaction with care measured by PASS-Opp | One year
  Satisfaction with care will be measured by PASS-Opp

CONTACTS AND LOCATIONS:
Overall Officials: Tore K Kvien, PhD, Study Director — Research director, Diakohjemmet Hospital
Locations (3):
- Norway (3):
  - Diakonhjemmet Hospital, Oslo
  - National resource center for rehabilitation in rheumatology, Oslo
  - Martina Hansens Hospital, Sandvika

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Polster A, Olsen U, Asphaug L, Bergsmark K, Christensen B, Haugen IK, Hennig T, Hermann-Eriksen M, Hove A, Sjovold T, Sexton J, Tveter AT, Kjeken I. Occupational therapist-led versus rheumatologist-led care in people with hand osteoarthritis in Norway: an open-label, multicentre, randomised controlled, non-inferiority trial. Lancet Rheumatol. 2025 Aug;7(8):e533-e543. doi: 10.1016/S2665-9913(25)00040-2. Epub 2025 Jun 10. PMID 40513596
- [Derived] Kjeken I, Bergsmark K, Haugen IK, Hennig T, Hermann-Eriksen M, Hornburg VT, Hove A, Proven A, Sjovold TA, Slatkowsky-Christensen B. Task shifting in the care for patients with hand osteoarthritis. Protocol for a randomized controlled non-inferiority trial. BMC Musculoskelet Disord. 2021 Feb 16;22(1):194. doi: 10.1186/s12891-021-04019-9. PMID 33593307
- See also: Published study protocol — https://pubmed.ncbi.nlm.nih.gov/33593307/

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-06-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03102788/SAP_001.pdf